CLINICAL TRIAL: NCT04782388
Title: A Placebo-Controlled, Double-blind, Randomized Study to Assess the Safety, Tolerability, And Pharmacokinetics of Staccato Alprazolam in Healthy Japanese, Chinese, and Caucasian Participants
Brief Title: Study to Assess the Safety, Tolerability, And Pharmacokinetics of Staccato Alprazolam in Healthy Japanese, Chinese, and Caucasian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UP0101
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Healthy Study Participants
Keywords: Healthy Study Participants; Phase 1; Staccato alprazolam; Alprazolam; STAP-001
MeSH Terms: interventions — Alprazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Staccato alprazolam (Experimental): Study participants will receive Single dose of Staccato alprazolam on Day 1 of the Treatment Period.
  Interventions: Drug: Alprazolam
- Staccato placebo (Placebo Comparator): Study participants will receive placebo on Day 1 of the Treatment Period.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Alprazolam — Study participants will receive Staccato alprazolam at prespecified time-point.
  Other Names: UCB7538
  Arms: Staccato alprazolam
Other: Placebo — Study participants will receive Staccato placebo at prespecified time-point.
  Other Names: PBO
  Arms: Staccato placebo

SUMMARY:
The purpose of the study is to assess the safety, tolerability, and pharmacokinetics (PK) of Staccato alprazolam in healthy Japanese, Chinese, and Caucasian participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent form (ICF)
* Participants are overtly healthy as determined by medical evaluation including medical history and physical examination
* For Japanese: Participant is of Japanese descent as evidenced by appearance and verbal confirmation of familial heritage (a participant has all 4 Japanese grandparents born in Japan) For Chinese: Participant is of Chinese descent as evidenced by appearance and verbal confirmation of familial heritage (a participant has all 4 Chinese grandparents born in China)
* Participant has a body weight (BW) of at least 45 kg (female) and 50 kg (male) and body mass index (BMI) within the range 18 to 30 kg/m^2(inclusive)

Exclusion Criteria:

* Participant has any medical or psychiatric condition that, in the opinion of the Investigator,could jeopardize or would compromise the study participant's ability to participate in this study
* Participant has a history or present condition of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders (eg, cardiac insufficiency, coronary heart disease, hypertension, arrhythmia, tachyarrhythmia, or myocardial infarction) capable of significantly altering the absorption, metabolism, or elimination of investigational medicinal product (IMP); constituting a risk when taking the study intervention; or interfering with the interpretation of data
* Participant has abnormal blood pressure (BP). Study participants must have BP and heart rate (HR) within normal range in the supine position after 5 minutes rest (systolic blood pressure (SBP): 90 mmHg to 140 mmHg, diastolic blood pressure (DBP): 50 mmHg to 90 mmHg, HR: 50 bpm to 100 bpm). Any values marginally (ie, no more than 5mmHg) outside the normal range but considered not clinically significant by the Investigator would be allowed. In case of an out-of-range result, 1 repeat will be allowed. If the readings are out of range again, the study participant will not be included
* Participant has a current history of alcohol or drug use disorder, as defined in Diagnostic and Statistical Manual of Mental Disorders V, within the previous 6 months
* Participant has a lifetime history of suicide attempt (including an actual attempt, interrupted attempt, or aborted attempt), or has had suicidal ideation in the past 6 months as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the "Screening/Baseline" version of the Columbia Suicide Severity Rating Scale (C-SSRS) at Screening
* Participant has history of or current clinical signs/symptoms consistent with suspected and/or confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)/coronavirus disease 2019 (COVID-19) (eg, fever, persistent cough, shortness of breath, fatigue, loss or change to senses of smell or taste)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Percentage of Japanese study participants with treatment-emergent adverse events (TEAEs) | From Baseline to the end of the Safety-Follow-Up (up to Day 10)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. The occurrence and incidence of TEAEs will also be summarized by intensity and by relationship to the investigational medicinal product (IMP).
Percentage of Japanese study participants with serious adverse event (SAEs) | From Baseline to the end of the Safety-Follow-Up (up to Day 10)
  A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose:
  1. Results in death
  2. Is life-threatening
  3. Requires inpatient hospitalization or prolongation of existing hospitalization
  4. Results in persistent disability/incapacity
  5. Is a congenital anomaly/birth defect
  6. Important medical events refered in the Protocol.
Percentage of Chinese study participants with treatment-emergent adverse events (TEAEs) | From Baseline to the end of the Safety-Follow-Up (up to Day 10)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. The occurrence and incidence of TEAEs will also be summarized by intensity and by relationship to the investigational medicinal product (IMP).
Percentage of Chinese study participants with serious adverse events (SAEs) | From Baseline to the end of the Safety-Follow-Up (up to Day 10)
  A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose:
  1. Results in death
  2. Is life-threatening
  3. Requires inpatient hospitalization or prolongation of existing hospitalization
  4. Results in persistent disability/incapacity
  5. Is a congenital anomaly/birth defect
  6. Important medical events refered in the Protocol.
Maximum plasma concentration (Cmax) of Staccato alprazolam in Japanese study participants | Plasma samples will be collected on predose within 30 minutes prior to dosing, at 1 minute, 2 minutes, 5 minutes, 10 minutes, and 30 minutes and at 1 hour, 2 hours, 4 hours, 6 hours, 12 hours, 24 hours, 36 hours, and 48 hours postdose
  Cmax = Maximum plasma concentration.
Area under the plasma concentration-time curve from time 0 to the last measurable concentration (AUClast) of Staccato alprazolam in Japanese study participants | Plasma samples will be collected on predose within 30 minutes prior to dosing, at 1 minute, 2 minutes, 5 minutes, 10 minutes, and 30 minutes and at 1 hour, 2 hours, 4 hours, 6 hours, 12 hours, 24 hours, 36 hours, and 48 hours postdose
  AUClast = Area under the plasma concentration-time curve from time 0 to the last measurable concentration.
Area under the plasma concentration-time curve from time 0 to infinity (AUCinf) of Staccato alprazolam in Japanese study participants | Plasma samples will be collected on predose within 30 minutes prior to dosing, at 1 minute, 2 minutes, 5 minutes, 10 minutes, and 30 minutes and at 1 hour, 2 hours, 4 hours, 6 hours, 12 hours, 24 hours, 36 hours, and 48 hours postdose
  AUCinf = Area under the plasma concentration-time curve from time 0 to infinity.
Maximum plasma concentration (Cmax) of Staccato alprazolam in Chinese study participants | Plasma samples will be collected on predose within 30 minutes prior to dosing, at 1 minute, 2 minutes, 5 minutes, 10 minutes, and 30 minutes and at 1 hour, 2 hours, 4 hours, 6 hours, 12 hours, 24 hours, 36 hours, and 48 hours postdose
  Cmax = Maximum plasma concentration.
Area under the plasma concentration-time curve from time 0 to the last measurable concentration (AUClast) of Staccato alprazolam in Chinese study participants | Plasma samples will be collected on predose within 30 minutes prior to dosing, at 1 minute, 2 minutes, 5 minutes, 10 minutes, and 30 minutes and at 1 hour, 2 hours, 4 hours, 6 hours, 12 hours, 24 hours, 36 hours, and 48 hours postdose
  AUClast = Area under the plasma concentration-time curve from time 0 to the last measurable concentration.
Area under the plasma concentration-time curve from time 0 to infinity (AUCinf) of Staccato alprazolam in Chinese study participants | Plasma samples will be collected on predose within 30 minutes prior to dosing, at 1 minute, 2 minutes, 5 minutes, 10 minutes, and 30 minutes and at 1 hour, 2 hours, 4 hours, 6 hours, 12 hours, 24 hours, 36 hours, and 48 hours postdose
  AUCinf = Area under the plasma concentration-time curve from time 0 to infinity.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of Staccato alprazolam in Caucasian study participants | Plasma samples will be collected on predose within 30 minutes prior to dosing, at 1 minute, 2 minutes, 5 minutes, 10 minutes, and 30 minutes and at 1 hour, 2 hours, 4 hours, 6 hours, 12 hours, 24 hours, 36 hours, and 48 hours postdose
  Cmax = Maximum plasma concentration.
Area under the plasma concentration-time curve from time 0 to the last measurable concentration (AUClast) of Staccato alprazolam in Caucasian study participants | Plasma samples will be collected on predose within 30 minutes prior to dosing, at 1 minute, 2 minutes, 5 minutes, 10 minutes, and 30 minutes and at 1 hour, 2 hours, 4 hours, 6 hours, 12 hours, 24 hours, 36 hours, and 48 hours postdose
  AUClast = Area under the plasma concentration-time curve from time 0 to the last measurable concentration.
Area under the plasma concentration-time curve from time 0 to infinity (AUCinf) of Staccato alprazolam in Caucasian study participants | Plasma samples will be collected on predose within 30 minutes prior to dosing, at 1 minute, 2 minutes, 5 minutes, 10 minutes, and 30 minutes and at 1 hour, 2 hours, 4 hours, 6 hours, 12 hours, 24 hours, 36 hours, and 48 hours postdose
  AUCinf = Area under the plasma concentration-time curve from time 0 to infinity.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- Up0101 101, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.